CLINICAL TRIAL: NCT01429753
Title: A Prospective Randomised Study of Advanced Imaging Guided Cardiac Resynchronisation Therapy (CRT) vs Conventional CRT Implantation in Patients With Chronic Heart Failure
Brief Title: PRISM Cardiac Resynchronisation Therapy (CRT) Randomised Controlled Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Manav Sohal, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0802/126
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Heart Failure
Keywords: Cardiac resychronisation therapy; Heart failure; Imaging guided LV lead placement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard LV lead placement (Active Comparator)
  Interventions: Device: Standard LV lead placement
- Advanced Imaging Guided LV Lead Placement (Experimental)
  Interventions: Other: Advanced Imaging Guided LV lead placement

INTERVENTIONS:
Other: Advanced Imaging Guided LV lead placement — Use of MRI to identify scar and latest activating LV segment as well as CS anatomy. This will be used to guide LV lead placement real-time.
  Arms: Advanced Imaging Guided LV Lead Placement
Device: Standard LV lead placement — Standard LV lead placement not guided by advanced imaging
  Arms: Standard LV lead placement

SUMMARY:
Cardiac resynchronisation therapy (CRT) is an established treatment for improving symptoms in patients with congestive heart failure (CHF) by left ventricular (LV) pacing. CRT can help to improve LV function in patients with heart failure if those regions of the myocardium which are most compromised by electromechanical dyssynchrony can be identified and effectively stimulated. There still remains, however, a significant rate of up to 30% of patients who do not respond to treatment. Reasons for lack of benefit can be related to the inability of identifying and effectively stimulating those regions of myocardium, which are most compromised by electromechanical dyssynchrony. The investigators hypothesize that by using cardiac MR and 3D echo to identify scar, reconstruct coronary sinus anatomy, and determine the site of latest LV activation, the investigators can find the best place to implant the left ventricular lead. By avoiding scar and pacing in the site of latest activation, the investigators believe the investigators will reduce dyssynchrony and thus improve overall heart function. The researchers thus aim to increase the proportion of people who respond to treatment. The researchers also believe that the procedure may be streamlined so as to reduce procedure duration, radiation dose and dose of iodinated contrast medium.

ELIGIBILITY:
Inclusion Criteria:

* >18yrs of age
* Standard indication for CRT=P or CRT=D according to NICE criteria (Clinical symptoms of heart failure despite medical therapy, broad QRS >120ms and significant LV dysfunction LEF <35%)
* Stable on optimal medical therapy for at least 3 months
* No exclusion to pacing /ICD
* Ischaemic or non-ischaemic aetiology

Exclusion Criteria:

* Any contraindication to pacing /ICD implant
* Contraindication to MR scanning
* Claustrophobia
* Significant renal impairment (estimated GFR <30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of CRT responders | 6 months

SECONDARY OUTCOMES:
Change in echo derived end systolic (ESV) and diastolic volumes | 6 months
Six month assessment of change in 6 minute walk distance and VO2 max (CPEX) | 6 months
Procedural success | 0 months
Procedure duration | 0 months
Radiation dose | 0 months
Contrast dose | 0 months
Procedural complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Aldo Rinaldi, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust